CLINICAL TRIAL: NCT06244706
Title: QSPainRelief-STRAT: A Questionnaire-based Evaluation of Perceived Clinical Outcome in Patients With Persistent Pain Receiving an Opioid and Non-opioid Treatment Combination, Stratified According to Age and Sex
Brief Title: QSPainRelief-STRAT
Acronym: QSPR-STRAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/13/JUI/259
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain; Analgesia; Adverse Drug Event; Drug Interaction
MeSH Terms: conditions — Chronic Pain; Agnosia; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peristent Pain Patients (Other): Patients suffering from persistent pain (pain lasting for at least three months), already treated with an opioid medication (treatment A) and to whom the treating physician is about to prescribe a CNS-acting add-on drug such as an antiepileptic, an antidepressant, a benzodiazepine or an alpha2-agonist (treatment B: the combination treatment), will be included.
  Evaluation of drug combination pain relief and its impact on daily life activities as therapeutic effects, and on drug-induced sedation and drug-induced cognitive dysfunction (memory and attention) as adverse effects will be evaluated through online (REDCap) patient-reported outcomes at the beginning of the study (day 0), 10 days and 3 months.
  Interventions: Combination Product: Opioid drug + CNS-acting add-on drug

INTERVENTIONS:
Combination Product: Opioid drug + CNS-acting add-on drug — Patients suffering from persistent pain (pain lasting for at least three months), already treated with an opioid medication (treatment A) and to whom the treating physician is about to prescribe a CNS-acting add-on drug such as an antiepileptic, an antidepressant, a benzodiazepine or an alpha2-agonist (treatment B: the combination treatment).

SUMMARY:
Investigating the clinical outcomes of drug combinations (opioid + medication acting on the central nervous system) in patients suffering from persistent pain (pain lasting for at least three months) through patient-reported outcomes.

DETAILED DESCRIPTION:
This study is part of the QSPainRelief project funded by the European Union's Horizon 2020 research and innovation program (grant agreement 848068; http://qspainrelief.eu).

The QSPainRelief project aims to setup, calibrate and validate a platform to predict the effects of treatment combinations according to patient characteristics such as age and sex (QSPainRelief platform) which integrates recently developed (1) physiologically based pharmacokinetic models to quantitate and adequately predict drug pharmacokinetics in human CNS, (2) target-binding kinetic models; (3) cellular signaling models and (4) a proprietary neural circuit model to quantitate the drug effects on the activity of relevant brain neuronal networks, that also adequately predicts clinical outcome.

To develop the QSPainrelief platform, a large dataset assessing perceived clinical outcome by real-world patients treated with a drug combination and stratified according to age and sex is required. To generate this dataset, we will conduct a questionnaire-based clinical study using an online platform (Redcap) and/or phone interviews to assess baseline patient characteristics and clinical outcome. Eligible patients are any patient treated with an opioid analgesic to whom an add-on treatment acting on the CNS is prescribed.

This study will focus on pain relief and its impact on daily life activities as therapeutic effects, and on drug-induced sedation, drug-induced cognitive dysfunction (memory and attention) and pain medication misuse as adverse effects. These adverse effects have been chosen because they can be readily assessed in patients after a short treatment period using validated patient-reported outcome measures (PROMs).

QSPainRelief-patientSTRAT is a monocentric prospective longitudinal questionnaire-based study conducted in patients suffering from persistent pain (pain lasting for at least three months), already treated with an opioid medication (treatment A) and to whom the treating physician is about to prescribe a CNS-acting add-on drug such as an antiepileptic, an antidepressant, a benzodiazepine or an alpha2-agonist (treatment B: the combination treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years.
2. Current treatment with an opioid for the treatment of pain, along with possible other drugs (see Table 1 for the list of eligible opioid medications - patients will be invited to indicate their treatment by selecting its name using a dropdown list).
3. Decision by the treating physician to introduce an additional non-opioid CNS-acting treatment such as an antiepileptic, an anti-depressant or benzodiazepine (see Table 2 for the list of eligible medications - patients will be invited to indicate their treatment by selecting its name using a dropdown list).
4. Capacity to understand and provide informed consent.

Exclusion Criteria:

1. Insufficient French language skills.
2. Epilepsy treated by an anti-epileptic.
3. Alzheimer's disease.
4. Parkinson's disease
5. History of cancer diagnosed less than 5 years ago, treated by chemotherapy or radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 10 days and 3 months
  The intensity of pain at 10 days and 3 months post-drug-combination compared vs. pre-drug combination. Assessment on how the combinational treatment influences pain relief, expressed as change in pain severity score from Day 0 to Day 10 and Month 3 realized with the Brief Pain Inventory (SF-BPI) pain severity score.
Daily Life Activities | 10 days and 3 months
  The impact on daily life activities at 10 days and 3 months post-drug combination compared vs. pre-drug combination. Assessment on how the combinational treatment influences daily activities, expressed as change in daily life activities score from Day 0 to Day 10, and Month 3, realized with the Brief Pain Inventory (SF-BPI) daily life activities score.
Quality of Life (EURO-QoL) | 3 months
  The impact on quality of life at 3 months post-drug-combination compared vs. pre-drug combination. Assessment on how the combinational treatment influences quality of life, expressed as change in EuroQOL-5D score from Day 0 to Month 3.
Drug-induced sedation | 10 days and 3 months
  Drug-induced sedation at 10 days and 3 months post-drug-combination compared vs. pre-drug combination. Assessment on how the combinational treatment influences sleepiness, expressed as change in the Stanford Sleepiness Scale score from Day 0 to Day 10 and Month 3
Drug-induced cognitive dysfunction | 10 days and 3 months
  . Drug-induced cognitive dysfunction (memory and attention) at 10 days and 3 months post-drug-combination compared vs. pre-drug combination. Assessment on how the combinational treatment influences cognitive functions, expressed as change in the PROMIS Neuro-QOL Short Form Cognitive Function score from Day 0 to Day 10 and Month 3.

IPD SHARING:
Plan to Share IPD: Undecided